CLINICAL TRIAL: NCT01655134
Title: Home-based Assessment of Plasma Volume, Serum Potassium and Renal Function Variations in Patients With Heart Failure and Low Left Ventricular Ejection Fraction: Pilot Study BIOMIC. Biomarkers and Therapeutic Modelisation in Heart Failure
Brief Title: Biomarkers and Therapeutic Modelisation in Heart Failure
Acronym: BIOMIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2012-A00306-37
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2013-07

CONDITIONS: Heart Failure
Keywords: Heart Failure; Telemonitoring systems for congestive HF; Biomarkers
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Blood simples
Other: Capillary punction
Other: Urine simples

SUMMARY:
The telemonitoring systems for congestive HF did not yet prove their efficacy despite initial encouraging results. Decongestion is one of the main objectives in Congestive HF, but an appropriate titration of diuretics is warranted, since long-term use of diuretics was consistently found associated with adverse outcomes. The investigators showed (ROSSIGNOL et al., JACC 2011, Circulation 2012) that the aldosterone antagonist eplerenone has diuretic effects, as assessed by an estimated plasma volume depletion, in addition to potassium-sparing properties, independently from renal function variations. These three parameters were independently associated with patient outcomes and may therefore be potential monitoring/and therapeutic targets in patients with congestive HF.

Main objective :

To assess the variations of estimated plasma volume, serum potassium and estimated glomerular filtration rate after an hospitalization for decompensated HF, by using a home-based finger capillary punction for 5 consecutive days per week during the two months postdischarge, using an approved dedicated device (ABOTT iSTAT).

Secondary objectives :

1. to assess the correlations between plasma volume, serum potassium and estimated glomerular filtration rate variations (as measured by Istat, and by a weekly venous punction) and body weight, home blood pressure measurement, dyspnea self assessment variations.
2. bio banking (serum, plasma, urine) for further biomarker studies, one a weekly basis

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or over
* Patients with heart failure and FE ≤ 45% hospitalized for decompensated heart failure

Exclusion Criteria:

* GFR < 30 ml/min/1.73 m2 as estimated by the abbreviated MDRD formula
* Pregnancy and lactation
* Participation in other investigational trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-01 (Estimated); Study Completion 2015-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Rossignol, Study Director — Brabois Hospital
Locations (1):
- Brabois hospital, Nancy, France

REFERENCES:
- [Derived] Rossignol P, Fay R, Girerd N, Zannad F. Daily home monitoring of potassium, creatinine, and estimated plasma volume in heart failure post-discharge. ESC Heart Fail. 2020 Jun;7(3):1257-1263. doi: 10.1002/ehf2.12642. Epub 2020 Apr 10. PMID 32274878